CLINICAL TRIAL: NCT01570127
Title: Clinical Trial to Evaluate and Compare the Efficacy and Safety of Individualized and Standardized Acupuncture for Low Back Pain Patients: Randomized, Double-blind, Controlled Study
Brief Title: Efficacy and Safety Study of Individualized and Standardized Acupuncture Treatment for Low Back Pain
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongwoo Nam (Other)
Collaborators: Ministry of Health & Welfare, Korea (Other Government); Gachon University Gil Medical Center (Other)
Responsible Party: Sponsor-Investigator, Dongwoo Nam, Assistant Professor, Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KOMCIRB-02-20101130-02
Record Dates: First submitted 2012-03-26; First posted 2012-04-04 (Estimated); Last update posted 2012-04-06 (Estimated); Status verified 2012-04

CONDITIONS: Low Back Pain
Keywords: Individualized Acupuncture; Standardized Acupuncture; Low Back Pain; Randomized Controlled Trial
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Individualized Acupuncture (Experimental): The patients in this group received individualized acupuncture prescribed by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 2 years of clinical experience. The acupuncture formulas were composed based on the pattern diagnosis, which is an unique diagnosis system of Oriental Medicine.
  Interventions: Procedure: Individualized Acupuncture
- Standardized Acupuncture (Experimental): The patients in this group received standardized acupuncture treatment using the same acupuncture points, applied by a certified Korean Medicine Doctor with more than 6 years of oriental medicine college education and 2 years of clinical experience. The acupuncture formulas were composed based on literature review of RCTs.
  Interventions: Procedure: Standardized Acupuncture
- Sham acupuncture (Sham Comparator): Non-penetrating acupuncture device, Park-sham acupuncture, was applied to the patients. The appearance of the acupuncture is same but the needles do not penetrate the skin.
  Interventions: Procedure: Sham Acupuncture
- Waiting (No Intervention): No interventions were applied to the patients in this group. Only assessments were made at each visit.
  Interventions: Other: Waiting

INTERVENTIONS:
Procedure: Individualized Acupuncture — The treatment was applied twice a week for 20 minutes for 6 weeks(12sessions)
  Arms: Individualized Acupuncture
Procedure: Standardized Acupuncture — The treatment was applied twice a week for 20 minutes for 6 weeks(12sessions) 8 Acupuncture points, GV4, GV3, BL24(bilateral), BL25(bilateral) and GB30(bilateral) were used for all the patients assigned to this group. Sterile Stainless Steel(25mm x 40mm) disposable acupuncture needles manufactured by Dong-Bang Acupuncture Co.(Korea) were used.
  Arms: Standardized Acupuncture
Procedure: Sham Acupuncture — The treatment was applied twice a week for 6 weeks(12sessions). The sham acupuncture was applied on the 8 same acupuncture points as in the standardized acupuncture group, GV4, GV3, BL24(bilateral), BL25(bilateral) and GB30(bilateral). Each session was 20 minutes long.
  Other Names: Park Sham Device
  Arms: Sham acupuncture
Other: Waiting — No interventions were applied to the patients in this group.
  Other Names: No interventions
  Arms: Waiting

SUMMARY:
The purpose of this study is to determine whether acupuncture treatment(Individualized & Standardized Acupuncture) is more effective than control (sham acupuncture or no treatment) and also whether individualized acupuncture is more effective than standardized acupuncture.

DETAILED DESCRIPTION:
To determine whether individualized acupuncture is more effective than standardized acupuncture, 276 Low Back Pain patients will be recruited and randomly assigned to 4 separate groups.

Experimental groups(Individualized Acupuncture Group and Standardized Acupuncture Group) and Control groups (Sham acupuncture and waiting list)

The change of pain and physical functions will be compared among the four groups.

So the efficacy of acupuncture, and the best acupuncture treatment model will be determined. Also in addition, safety and abnormal reactions of acupuncture treatments will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients suffering Low Back Pain.
* Patients classified as Class 1(pain in the lumbar area, without radiation below the gluteal fold and in the absence of neurologic signs) or Class 2(Low back pain with radiation of pain not beyond the knee, no neurological signs) according to the Quebec Task Force System
* Suffering pain which is more than 40mm on VAS(Visual Analog Scale)
* Voluntary participants who have completed the consent.

Exclusion Criteria:

* Low back trauma history within 6 months.
* Low back surgery history within 6 months.
* Low back pain caused by malignancy, inflammatory disease, fibromyalgia, vertebral fracture, infection, juvenile scoliosis or congenital malformation.
* Pain in other parts of the body more severe than low back pain.
* Mental problems that can influence the pain or results of questionnaire.
* Diseases that can interfere absorption, metabolism and excretion of medicine.
* History of alcohol or drug abuse within 12 months of the study.
* Pregnant, breastfeeding or childbearing aged women who are not using any birth control methods.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2010-10; Primary Completion 2012-08 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
The change of 100mm pain Visual Analog Scale(VAS) after 6 weeks of treatment. | at baseline and after 6 weeks of treatment.
  Visual analog scale (VAS) is a tool used to measure pain. The patient is asked to indicate their perceived pain intensity along a 100 mm horizontal line, where '0' represents 'no pain' and '100', 'unbearable pain'. The change of pain will be reported by comparing the mean VAS before treatment and after the 6 week trearment period.

SECONDARY OUTCOMES:
Roland - Morris Disability Questionnaire | at 2nd(baseline), 8th(after 4 weeks of treatment), 13th(end of study) and 14th(follow up) visit
  Roland - Morris Disability Questionnaire (RMDQ) is scored by adding up the number of items checked by the patients, among the 24 items concerning various disablilities caused by low back pain. The score can therefore vary from 0 to 24. Higher the scores represent worse disabilities.
SF-36 | at 2nd(baseline), 8th(after 4 weeks of treatment), 13th(end of study) and 14th(follow up) visit
  The 36 questions yields an 8-scale health profile. It is useful in monitoring the change in health related quality of life.
Adverse Events | at 2nd(baseline), 3rd, 4th, 5th, 6th, 7th, 8th, 9th, 10th, 11th, 12th and 13th(end of study)
  Any unpredicted symptoms were checked at each follow up visit and if any, the symptom, time of occurrence, and length of duration were recorded and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Dong Lee, Ph.D, Study Chair — Kyunghee University Medical Center
Locations (1):
- Kyung Hee University Oriental Medicine Hospital, Seoul, Seoul, South Korea